CLINICAL TRIAL: NCT03071744
Title: Phase II, Open-Label Study to Evaluate Lazanda in Cancer Patients Receiving Palliative Radiation
Brief Title: Lazanda in Cancer Patients Receiving Palliative Radiation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI is leaving UCSD
Sponsor: Joseph Ma (Other)
Responsible Party: Sponsor-Investigator, Joseph Ma, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCSD 161263
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Results first posted 2019-07-23 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lazanda (Other): Study drug, Lazanda, will be self-administered intranasally during this study. The dose of Lazanda is not predicted from the daily maintenance dose of opioid used to manage persistent cancer pain and must be determined by dose titration. The minimal effective intranasal dose from the radiation therapy simulation will be the dose used as pre-medication prior to any further radiation therapy fractions (up to 10 fractions).
  Lazanda should be administered 15 (T-15) minutes prior to laying on the hard surface for each simulation visit. If the response to the titrated Lazanda dose markedly changes, an adjustment of dose may be necessary to ensure that an appropriate dose is maintained as deemed by the investigator.
  Interventions: Drug: Lazanda

INTERVENTIONS:
Drug: Lazanda — Lazanda is supplied in glass bottles, containing 8 sprays of 100 mcL containing 100 mcg/100 mcL or 400 mcg/100 mcL concentration solution.
  Other Names: Fentanyl

SUMMARY:
Advanced cancer patients often require palliative (pain relieving) radiotherapy to treat cancer-related symptoms. The delivery of radiation requires patients to lie still on a hard flat surface, which can result in significant acute (intense) pain and/or breakthrough cancer pain (sudden sharp or stabbing pain), especially when painful bone metastases are present. The current care for most cancer patients receiving radiation is to take an oral (by mouth) opioid medication before the radiation treatment. The pain relieving effects of these medications can take about one hour and can last for 3 to 6 hours, which does not follow the time course of when breakthrough cancer pain occurs.

Lazanda is a pain medication delivered via an intranasal route and is already approved by the U.S. Food and Drug Administration (FDA) for the management of breakthrough cancer pain for patients who are already receiving opioids and who can tolerate opioids for the treatment of cancer pain. Lazanda is fast-acting and convenient for patients to take. The purpose of this study is to assess the change in pain intensity during palliative radiotherapy following study treatment with Lazanda. This study will also explore the impact of the study treatment on the efficiency in delivering the radiation therapy

DETAILED DESCRIPTION:
This is a Phase II, single-center, single-arm, Open-Label Study to Evaluate Lazanda in Cancer Patients Receiving Palliative Radiation.

The primary objective of this study is to assess the change in patient reported positional pain intensity (PI) as measured by an 11-point numerical rating scale (NRS-11) in cancer patients with bone metastases assessed at a simulation visit and each subsequent daily palliative radiation fraction. The primary objective will be measured using the pain intensity difference (PID) of the NRS-11 from the time of laying down on the hard surface (0 minutes/ PI0) to the 15 minutes after laying down on the hard surface timepoint at baseline (the simulation visit) and at each subsequent study visit (PID15= PI0- PI15).

Study participants will be recruited across all oncology disease teams. Potential participants will be identified in weekly palliative care or disease team patient triage meetings. In order to meet eligibility for participation, a patient must be greater than or equal to 18 years old, have histologically-confirmed cancer with symptomatic bone metastases, an Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 3, and are planned to receive hypofractionated palliative radiation less than or equal to 10 fractions. Qualifying subjects must be opioid-tolerant, defined as greater than or equal to 60mg morphine or equivalent, and be on a stable dose of oral opioids for greater than or equal to 1 week. Stable baseline opioid dosage is defined as a dosage that does not fluctuate by more than 50% from the average dosage over one week prior to screening. Patients must also be on a stable dose of adjuvant pain therapies for one week prior to screening. Patients will be excluded if they are receiving or have received another investigational agent within 30 days or monoamine oxidase inhibitor within 14 days prior to Lazanda administration, have known hypersensitivity to fentanyl or opioids, have known, planned interventional procedures such as surgery that may affect study outcomes, are pregnant or nursing, have a disorder or current medication use likely to adversely affect normal functioning of the nasal mucosa, have uncontrolled or rapidly escalating background pain, or are medically unstable, require immobilization with a thermoplastic mask for radiation treatment.

Upon confirmation of all eligibility criteria, the subject will be enrolled. Each enrolled subject will undergo a baseline evaluation on a mock hard surface within 1 week prior to the time of CT simulation, to establish baseline NRS pain scores.

Subject will receive Lazanda at their mock hard surface visit , radiation simulation visit and again as pre-medication prior to each radiation treatment (fraction), for an estimated treatment period of 10 days based on the patient's radiation treatment plan. Lazanda will be self-administered intranasally by subjects participating in this study.

NRS pain scores will be collected at three time points at baseline : 15 minutes prior to laying on the hard surface (T-15), at the time of laying on the hard surface (T0), and at 15 minutes after laying on the hard surface(T+15). Exact time of each pain score rating will also be collected.

After the mock visit subject will then undergo radiation therapy simulation procedures (within approximately 2 weeks of radiation therapy) followed by hypofractionated radiation therapy, according to University of California, San Diego (UCSD) Radiation Oncology standard procedure and treatment plan determined by the subject's radiation oncologist. During radiation simulation and daily during each visit to the radiation center for hypofractionation delivery, subjects will have vital signs and weight collected. An ECOG performance status will also be assessed daily during radiation therapy. At the time of radiation simulation and daily during radiation therapy, subjects will complete the BPI-sf , Medication Use Diary, Laxation Diary, and Nausea/Vomiting Diary. As with the mock hard surface evaluation, NRS pain scores will also be collected at three time points during each visit to the radiation center.

Subjects will receive study drug, Lazanda at 100mcg dose, 15 minutes prior to simulation (T-15) at the radiation therapy simulation visit. Lazanda dose titration will follow the guidelines as indicated in the product package insert from the radiation simulation visit through the end of radiation therapy.

Subjects will undergo a post treatment follow-up period after completion of their radiation therapy. During this follow-up period, subjects will complete the BPI-sf, Medication Use Diary, Laxation Diary , and Nausea/Vomiting Diary daily for 2 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has the ability to understand and the willingness to sign a written informed consent.
2. Pathologically-confirmed solid tumor or hematologic malignancy with symptomatic bone metastases.
3. Patient is planned to receive hypofractionated palliative radiation ≤ 10 fractions.
4. Patient must be opioid-tolerant (greater than or equal to 60mg morphine or equivalent) and on a stable dose of oral opioids for greater than or equal to 1 week. Stable baseline opioid dosage defined as a dosage that does not fluctuate by more than 50% from the average dosage over one week prior to screening.
5. Patient must be on a stable dose of adjuvant pain therapies for one week prior to screening (i.e. steroids, NSAIDs, anticonvulsants, pharmaceutical cannabinoids, tricyclic antidepressants).
6. Patient is ≥ 18 years of age.
7. Both men and women of all races and ethnic groups are eligible for this trial.
8. ECOG Performance Status ≤ 3
9. Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 28 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

   * A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
10. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)Women of child-bearing potential has negative pregnancy test prior to initiating study drug dosing.

Exclusion Criteria:

1. Patient is currently receiving or has received another investigational agent within 30 days or monoamine oxidase inhibitor within 14 days prior to Lazanda administration.
2. Patients who require immobilization with a thermoplastic mask for radiation treatment.
3. Patient is planned to receive interventional procedures (i.e. surgery) that may affect study outcomes.
4. Patient has a history of hypersensitivity to fentanyl or opioids.
5. Patient is pregnant or nursing. There is a potential for congenital abnormalities and for this regimen to harm nursing infants.
6. Patient is being treated with oxymetazoline for allergic rhinitis or has a disorder or current medication use likely to adversely affect normal functioning of the nasal mucosa.
7. Patient has uncontrolled or rapidly escalating background pain.
8. Patient has bradyarrhythmia.
9. Patient is considered medically unstable.
10. Patient is thought to be at risk for misuse, abuse, addiction or overdose for Schedule II controlled substance, as evidenced by the following:

    1. An Opioid Risk Tool (ORT) score of greater/less than or equal to 8.
    2. A review of the California Prescription Control Monitoring Program (PDMP) Controlled Substance Utilization Review and Evaluation System (CURES) report demonstrates multiple prescribing providers and/or multiple pharmacies in the last 30 days. The CURES report will also be used to verify opioid use, opioid dose, and current prescribing providers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ma, PharmD, Principal Investigator — UCSD
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lazanda: Study drug, Lazanda, will be self-administered intranasally during this study. The dose of Lazanda is not predicted from the daily maintenance dose of opioid used to manage persistent cancer pain and must be determined by dose titration. The minimal effective intranasal dose from the radiation therapy simulation will be the dose used as pre-medication prior to any further radiation therapy fractions (up to 10 fractions).
  Lazanda should be administered 15 (T-15) minutes prior to laying on the hard surface for each simulation visit. If the response to the titrated Lazanda dose markedly changes, an adjustment of dose may be necessary to ensure that an appropriate dose is maintained as deemed by the investigator.
  Lazanda: Lazanda is supplied in glass bottles, containing 8 sprays of 100 mcL containing 100 mcg/100 mcL or 400 mcg/100 mcL concentration solution.
Period: Overall Study
Arm/Group | Lazanda
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lazanda
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Patient Reported Positional Pain Intensity
Description: Assess the change in patient reported positional pain intensity (PI) as measured by an 11-point numerical rating scale zero (no pain) to ten (severe pain) (NRS-11; scores on a scale) in cancer patients with bone metastases assessed at each daily palliative radiation fraction. Our primary objective will be measured using the pain intensity difference (PID) of the NRS-11 between 0 minutes and 15 minutes after laying down on the hard surface (PID15= PI0- PI15).
Time Frame: 0 minutes and 15 minutes after laying down on the hard surface (PID15= PI0- PI15).
Measure: Count of Participants; unit: Participants
Arm/Group | Lazanda
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Participants With Change in Patient Reported Positional Pain Severity Via the Brief Pain Inventory Short Form
Description: Assess change in patient reported pain severity using the Brief Pain Inventory Short Form (BPI-sf).
Time Frame: from the time of laying down on the hard surface (0 minutes) to 15 minutes after laying down at each fractionation visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Lazanda
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Number of Participants With Adverse Effects Associated With Lazanda
Description: evaluate adverse effects associated with Lazanda use utilizing the NCI CTCAE version 4.03 before and after palliative radiation.
Time Frame: 4-5 weeks of patient participation in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Lazanda
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 30 days from the last study drug administration (about 2 months)
Arm/Group | Lazanda
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lazanda (N=6)
Sepsis due to UTI (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lazanda (N=6)
Dry Heaves (Gastrointestinal disorders) | 1
Malaise - aches /pain (Musculoskeletal and connective tissue disorders) | 1
Flu Symptoms (Immune system disorders) | 1
Severe leg pain (Musculoskeletal and connective tissue disorders) | 1
Dry mouth (Skin and subcutaneous tissue disorders) | 1
Creatinine increase (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT03071744/Prot_SAP_000.pdf